CLINICAL TRIAL: NCT06952270
Title: Effects of Two Strength Exercise Programs on Upper Limb Functionality in Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Yoana González González, Principal Investigator, University of Vigo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28022025
Record Dates: First submitted 2025-03-29; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Survivor; Breast Cancer; Breast Cancer Patients; Breast Cancer - Female
Keywords: breast cancer; plyometric exercise; upper limb; strength training; exercise; Recovery of Function; clinical trial
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- plyometric exercise group (Experimental): this group will perform a program of different exercises focused on the upper limb and shoulder girdle based on plyometric exercises.
  Interventions: Other: plyometric exercise
- Strength training exercise group (Experimental): This group will perform a strength training program by performing different exercises focused on the upper limb, lower limb and trunk muscle strengthening.
  Interventions: Other: Strength training exercise

INTERVENTIONS:
Other: plyometric exercise — Upper limb plyometric exercise (proprioceptive neuromuscular facilitation of extensor and flexor pattern, external rotation exercise at 90º-90º, chest throw, external rotation and overhead and wall flexion).
  Arms: plyometric exercise group
Other: Strength training exercise — Strength training exercises (Squats, Stair climbing and jumps, Bench Press, Push-ups, Core Exercises (Plank, Bridge)).
  Arms: Strength training exercise group

SUMMARY:
The goal of this experimental study is to evaluate the effect of a therapeutic exercise program based on upper limb plyometric exercises in breast cancer patients and breast cancer survivors to determine changes in upper limb functionality.

The main question it aims to answer is: Does upper limb plyometric strength exercise improve upper limb dysfunctions in breast cancer patients and survivors? The researchers will compare the effects of plyometric exercise with the effects of strength training exercise to determine whether plyometric exercise improves shoulder dysfunctions in breast cancer patients and survivors.

Participants from the Pontevedra group will undergo the intervention using plyometric exercise (Experimental Group), while those from the Vigo group will perform strength training exercise (Control Group). They will complete two sessions per week for six weeks. Outcome variables related to upper limb functionality will be assessed at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of breast cancer.
* Patients who have undergone a mastectomy, including unilateral, total breast, or breast-conserving surgery.
* Postoperative chemotherapy or radiotherapy as required.
* No other malignant tumors in the last 5 years.
* Absence of contraindications related to physiotherapy or physical exercise.
* Willingness to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Metastasis to other organs and tissues (liver, kidney, lung, brain, etc.) that prevent participation in the exercise program.
* Underlying heart disease, cerebrovascular disease, or mental illness that impairs proper execution of the exercise program.
* Pre-existing shoulder pathology before surgery.
* Inability to understand the plyometric exercise program.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in pain and activities of daily living, range of motion in flexion, abduction, external rotation, and internal rotation and sustained submaximal strength at six weeks | From enrollment to the end of treatment at 6 weeks
  Constant-Murley Score (Spanish version):
  Minimum and maximum values: 0 to 100. The scoring system includes 35 points for subjective measurement and 65 points for objective measurement.
  Interpretation: Higher scores indicate less disability.
Change from Baseline in Disability Arm Shoulder and Hand at six weeks | From enrollment to the end of treatment at 6 weeks
  Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire:
  Minimum and maximum values: The Spanish version of the DASH is a 30-item questionnaire where each question offers response options ranging from "no difficulty" or "none," scored as 1, to "unable" or "very severe," scored as 5. The total score ranges from 0 (no disability) to 100 (severe disability). At least 27 out of 30 questions must be completed to calculate a score. The values assigned to each response are summed and divided by the number of responses to obtain an average score from 1 to 5. This value is then transformed to a 0-100 score by subtracting 1 and multiplying by 25. This transformation facilitates comparison with other tools that report results on a 0-100 scale.
  Interpretation: Higher scores indicate greater disability.
Change from baseline in the maximum grip muscle strength at six weeks | "From enrollment to the end of treatment at 6 weeks"
  Minimum and maximum values: Maximum grip strength is measured using dynamometry and determined by the average of three measurements at each time point.
  Interpretation: Higher scores indicate less disability.
Change from baseline in the proprioception at six weeks | "From enrollment to the end of treatment at 6 weeks"
  Assessed by determining force sense: First, maximum grip strength is measured, and the participant is then asked to reproduce half of that maximum force. Three measurements are taken, and the one closest to the target is recorded.
  Additionally, proprioception is assessed by determining joint position sense (statesthesia): The examiner moves the subject's wrist, and the subject is asked to memorize the position to reproduce it later with their eyes closed. In a second phase, with eyes covered, the subject is asked to reach the previously indicated position from a starting point. Any deviation from the neutral position is measured using a goniometer. One measurement is taken for each position, and the closest one is recorded.
Change from baseline in the maximum isometric upper limb strength at six weeks | "From enrollment to the end of treatment at 6 weeks"
  The variable of maximum isometric upper limb strength will be measured using the MicroFET2 in internal rotation, external rotation, and flexion, all performed in the scapular plane. Two measurements of maximum strength will be taken, with 30 seconds of rest between attempts. Each contraction will be held for 3 seconds.
  The researcher will passively position the upper limb at 0º of shoulder flexion and 90º of elbow flexion, with the force applied to the palmar side of the distal third of the forearm for internal rotation, and to the dorsal side for external rotation. For flexion, the arm will be positioned at 90º of shoulder flexion in the scapular plane and 90º of elbow flexion, with force applied at the distal part of the humerus.
  Minimum and maximum values: The test is performed twice, and the highest value is recorded.
  Interpretation: Higher scores indicate better results.
Change from baseline in the circumference measurement: at six weeks | "From enrollment to the end of treatment at 6 weeks"
  The diameter of the upper limb with lymphedema will be measured using a thin, flexible plastic measuring tape at four anatomical points: the metacarpophalangeal joint, the wrist, 10 cm below, and 10 cm above the lateral epicondyles. The subject will be positioned in a supine position with the arm in the anatomical position, in supination. Three measurements will be taken at each point, and the average of the three measurements will be calculated.
Change from baseline in the kinesiophobia at six weeks | "From enrollment to the end of treatment at 6 weeks"
  Tampa Scale of Kinesiophobia-11 (TSK-11): The score ranges from 11 to 44. Interpretation: The lowest score (11) indicates no or insignificant kinesiophobia, and higher scores indicate increasing levels of kinesiophobia.
Change from baseline in the Sensation of heaviness of the upper limb at six weeks | From enrollment to the end of treatment at 6 weeks
  Minimum and maximum values: The reported value is recorded using a visual analog scale from 0 to 10, where 0 means no heaviness and 10 means maximum heaviness.
  Interpretation: Higher scores indicate greater disability.
Change from baseline in the Sensation of pain of the upper limb at six weeks | From enrollment to the end of treatment at 6 weeks
  Minimum and maximum values: The reported value is recorded using a visual analog scale from 0 to 10, where 0 means no pain and 10 means maximum pain.
  Interpretation: Higher scores indicate greater disability.
Change from baseline in the Sensation of tension of the upper limb at six weeks | From enrollment to the end of treatment at 6 weeks
  Minimum and maximum values: The reported value is recorded using a visual analog scale from 0 to 10, where 0 means no tension and 10 means maximum tension.
  Interpretation: Higher scores indicate greater disability.

SECONDARY OUTCOMES:
Sex | At the baseline
  Female
Age | At the baseline
  Years
Weight | At the baseline
  Kilograms (measured using a Tanita electronic scale [model 780 MA portable]; with a measurement range of 0-200 kg and d=0.1 kg)
Height | At the baseline
  Centimeters (measured using a stadiometer, d=0.1 mm and measurement range of 0 to 2000 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy of Pontevedra, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin Y, Wu C, He C, Yan J, Chen Y, Gao L, Liu R, Cao B. Effectiveness of three exercise programs and intensive follow-up in improving quality of life, pain, and lymphedema among breast cancer survivors: a randomized, controlled 6-month trial. Support Care Cancer. 2022 Dec 13;31(1):9. doi: 10.1007/s00520-022-07494-5. PMID 36512157
- [Background] Shao YW, Shu Q, Xu D, Teng H, Wu GS, Hou JX, Tian J. Effect of different rehabilitation training timelines to prevent shoulder dysfunction among postoperative breast cancer patients: study protocol for a randomized controlled trial. Trials. 2021 Jan 6;22(1):16. doi: 10.1186/s13063-020-04954-3. PMID 33407753
- [Background] Hasenoehrl T, Palma S, Ramazanova D, Kolbl H, Dorner TE, Keilani M, Crevenna R. Resistance exercise and breast cancer-related lymphedema-a systematic review update and meta-analysis. Support Care Cancer. 2020 Aug;28(8):3593-3603. doi: 10.1007/s00520-020-05521-x. Epub 2020 May 15. PMID 32415386
- [Background] Swanik KA, Thomas SJ, Struminger AH, Bliven KC, Kelly JD, Swanik CB. The Effect of Shoulder Plyometric Training on Amortization Time and Upper-Extremity Kinematics. J Sport Rehabil. 2016 Dec;25(4):315-323. doi: 10.1123/jsr.2015-0005. Epub 2016 Aug 24. PMID 27632848